CLINICAL TRIAL: NCT01213680
Title: Open-label Pharmakokinetic Study of Iron Isomaltoside 1000 (Monofer)Administered by 500 mg IV Injection or 1000 mg Intravenous Infusion to Patients With Inflammatory Bowel Disease (PK-IBD-02)
Brief Title: Open-label PK Study of Iron Isomaltoside 1000 (Monofer) Administered by 500 mg IV Injection or 1000 mg IV Infusion to Patients With Inflammatory Bowel Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-Monofer-PK-IBD-02; PK-IBD-02
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Inflammatory Bowel Disease
Keywords: Inflammatory Bowel Disease, IBD
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — iron isomaltoside 1000

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1000 mg iron isomaltoside as intravenous infusion (Active Comparator)
  Interventions: Drug: Monofer (iron isomaltoside 1000)
- 500 mg iron isomaltoside 1000 as bolus injection (Active Comparator)
  Interventions: Drug: Monofer

INTERVENTIONS:
Drug: Monofer (iron isomaltoside 1000) — 1000 mg iron isomaltoside administered as a infusion over 15 minutes
  Arms: 1000 mg iron isomaltoside as intravenous infusion
Drug: Monofer — 500 mg iron isomaltoside 1000 given as bolus injection over 2 minutes
  Arms: 500 mg iron isomaltoside 1000 as bolus injection

SUMMARY:
The purpose of this study is to assess the pharmakokinetic properties of higher doses (500 mg and 1000 mg) of Monofer(R)in patients suffering from inflammatory bowel disease

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged more than 18 years
2. Subjects diagnosed with inflammatory bowel disease and mild to moderate disease activity (defined as a score of less than or equal to 5 on the Harvey-Bradshaw index for Crohn's disease and a Mayo score (subscore without endoscopy) of less than or equal to 6 for ulcerative colitis)
3. Weight above 50 kg
4. Hb <12 g/dL (7.45 mmol/L)
5. Transferrin saturation (TfS) <20%
6. Life expectancy beyond 12 months by investigator's judgment
7. Willingness to participate after informed consent -

Exclusion Criteria:

1. Anaemia predominantly caused by other factors than iron deficiency anaemia
2. Iron overload or disturbances in utilisation of iron (e.g. haemochromatosis and haemosiderosis)
3. Drug hypersensitivity (i.e. previous hypersensitivity to Iron Dextran or iron mono- or disaccharide complexes or to iron sulphate)
4. Known hypersensitivity to any excipients in the investigational drug products
5. Subjects with a history of multiple allergies
6. Active Intestinal Tuberculosis
7. Active intestinal amoebic infections
8. Decompensated liver cirrhosis and hepatitis (Alanine Aminotransferase (ALT) > 3 times upper limit normal)
9. History of immunocompromise and/or history of Hepatitis B and/or C
10. Acute infections (assessed by clinical judgment), supported by white blood cells (WBC) and C-reactive protein (CRP))
11. Rheumatoid arthritis with symptoms or signs of active joint inflammation
12. Pregnancy and nursing (To avoid pregnancy, women have to be postmenopausal (at least 12 months must have elapsed since last menstruation), surgically sterile, or women of child bearing potential must use one of the following contraceptives during the whole study period and after the study has ended for at least 5 times plasma biological half-life of the investigational medicinal product: Contraceptive pills, intrauterine devices (IUD), contraceptive depot injections (prolonged-release gestagen), subdermal implantation, vaginal ring, and transdermal patches)
13. Extensive active bleeding necessitating blood transfusion
14. Planned elective surgery during the study
15. Participation in any other clinical study within 3 months prior to screening
16. Untreated B12 or folate deficiency
17. Other I.V. or oral iron treatment or blood transfusion within 4 weeks prior to screening visit
18. Erythropoietin treatment within 4 weeks prior to screening visit
19. Any other medical condition that, in the opinion of Investigator, may cause the patient to be unsuitable for the completion of the study or place the patient at potential risk from being in the study. Example: Uncontrolled Hypertension, Unstable Ischemic Heart Disease or Uncontrolled Diabetes Mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-02; Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Total serum iron pharmakokinetic parameters | 24, 48 and72 hours

SECONDARY OUTCOMES:
Total urine-iron pharmakokinetic parameters | 24, 48 and 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Lars Lykke Thomsen, MD, Study Chair — Pharmacosmos A/S